CLINICAL TRIAL: NCT00243659
Title: An Open Label Multi-center Study to Assess the Efficacy and Safety of B-Domain Deleted Recombinant Factor VIII (BDDrFVIII, ReFacto AF) in Patients With Hemophilia A Undergoing Elective Major Surgery
Brief Title: Study Evaluating B-Domain Deleted Recombinant Factor VIII (BDDrFVIII, ReFacto AF) in Patients With Hemophilia A Undergoing Elective Major Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-311
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; bleeding disorder
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders | interventions — Factor VIII

ARMS (2):
- A (Experimental)
  Interventions: Biological: ReFacto AF
- B (Experimental)
  Interventions: Biological: ReFacto AF

INTERVENTIONS:
Biological: ReFacto AF

SUMMARY:
This study will examine the efficacy and safety of ReFacto AF in patients with severe and moderately severe hemophilia A undergoing elective major surgery when administered by either bolus injections (BI) or continuous infusion (CI).

ELIGIBILITY:
* Male, at least 12 years old, with severe hemophilia A undergoing major elective major surgery requiring FVIII replacement for at least 6 days. Negative FVIII inhibitor test at screening and no past history of inhibitor.
* Previously treated with at least 150 exposure days to any Factor VIII product
* Normal hepatic and renal function tests and no other bleeding disorder

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (16):
- United States (7):
  - La Jolla, California
  - Detroit, Michigan
  - Chapel Hill, North Carolina
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Charlottesville, Virginia
- Perth, Australia
- Vienna, Austria
- Budapest, Hungary
- New Zealand (2):
  - Auckland
  - Chirstchurch
- Warsaw, Poland
- Bucurest, Romania
- Sweden (2):
  - Malmo
  - Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from April 2006 to April 2008.
Pre-assignment Details: Patients were screened for a maximum of 42 days.
Groups:
- Bolus Injection: Approximately 50 IU/kg Refacto AF for 6 consecutive days
- Continuous Infusion: Approximately 50 IU/Kg Refacto AF then continuously
Period: Overall Study
Arm/Group | Bolus Injection | Continuous Infusion
Started | 22 | 8
Completed | 20 | 5
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bolus Injection | Continuous Infusion | Total
Number analyzed (Participants) | 22 | 8 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 35.05 (9.51) | 38.13 (8.54) | 35.87 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0.0
  Male | 22 | 8 | 30.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Hemostatic Efficacy After Surgery
Description: Efficacy at the end of surgery as determined by the investigator and/or the surgeon using the 4 point ordinal scale (Excellent, Good, Moderate or None). Excellent: Achieved hemostatic comparable to non-hemophilic patients. Good: Prolonged time to hemostasis (with somewhat increased bleeding compared to non-hemophilic patients.
Time Frame: 6 weeks
Population: The analysis population is the efficacy evaluable at visit three.
Measure: Number; unit: patients
Arm/Group | Bolus Injection | Continuous Infusion
Number analyzed (Participants) | 20 | 5
patients
  Excellent | 15 | 3
  Good | 5 | 2
  Moderate | 0 | 0
  None | 0 | 0

2. Secondary Outcome: Number of Patients Who Achieved Hemostatic Efficacy at Hospital Discharge
Description: Assessment of hemostatic efficacy by the investigator at the day of discharge from the hospital using the 4 point ordinal scale (Excellent, Good, Moderate or None). Excellent: Achieved hemostatic comparable to non-hemophilic patients. Good: Prolonged time to hemostasis (with somewhat increased bleeding compared to non-hemophilic patients.
Time Frame: 6 weeks
Population: The analysis population is the efficacy evaluable at visit five.
Measure: Number; unit: patients
Arm/Group | Bolus Injection | Continuous Infusion
Number analyzed (Participants) | 20 | 5
patients
  Excellent | 18 | 5
  Good | 2 | 0
  Moderate | 0 | 0
  None | 0 | 0

ADVERSE EVENTS:
Arm/Group | Bolus Injection | Continuous Infusion
Serious Adverse Events (participants affected / at risk) | 4 | 1
Other Adverse Events (participants affected / at risk) | 19 | 7
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Bolus Injection | Continuous Infusion
Fever (General disorders) | 0/22 | 1/8
Accidental injury (General disorders) | 1/22 | 0/8
Cellulitis (General disorders) | 1/22 | 0/8
Hemorrhage (Cardiac disorders) | 0/22 | 1/8
Factor VIII inhibition (Blood and lymphatic system disorders) | 2/22 | 0/8
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0/22 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Bolus Injection | Continuous Infusion
Accidental injury (General disorders) | 3/22 | 0/8
Asthenia (General disorders) | 0/22 | 1/8
Back pain (General disorders) | 1/22 | 0/8
Cellulitis (General disorders) | 1/22 | 0/8
Chills (General disorders) | 2/22 | 0/8
Fever (General disorders) | 7/22 | 6/8
Flu syndrome (General disorders) | 3/22 | 0/8
Headache (General disorders) | 3/22 | 1/8
Injection (General disorders) | 5/22 | 0/8
Non-specified drug reaction (General disorders) | 0/22 | 1/8
Pain (General disorders) | 2/22 | 6/8
Hemorrhage (Cardiac disorders) | 0/22 | 1/8
Hypertension (Cardiac disorders) | 2/22 | 1/8
Hypotension (Cardiac disorders) | 1/22 | 0/8
Hypovolemia (Cardiac disorders) | 0/22 | 1/8
Pallor (Cardiac disorders) | 0/22 | 1/8
Tachycardia (Cardiac disorders) | 0/22 | 1/8
Abdominal distension (Gastrointestinal disorders) | 0/22 | 1/8
Constipation (Gastrointestinal disorders) | 1/22 | 0/8
Diarrhea (Gastrointestinal disorders) | 1/22 | 0/8
Jaundice (Gastrointestinal disorders) | 0/22 | 1/8
Mouth ulceration (Gastrointestinal disorders) | 1/22 | 0/8
Nausea (Gastrointestinal disorders) | 3/22 | 1/8
Vomiting (Gastrointestinal disorders) | 1/22 | 1/8
Anemia (Blood and lymphatic system disorders) | 8/22 | 1/8
Leukocytosis (Blood and lymphatic system disorders) | 0/22 | 1/8
Thrombocythemia (Blood and lymphatic system disorders) | 2/22 | 1/8
Bilirubinemia (Metabolism and nutrition disorders) | 0/22 | 1/8
Peripheral edema (Metabolism and nutrition disorders) | 1/22 | 1/8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/22 | 0/8
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1/22 | 0/8
Hypesthesia (Nervous system disorders) | 1/22 | 0/8
Memory impairment (Nervous system disorders) | 0/22 | 1/8
Paresthesia (Nervous system disorders) | 1/22 | 0/8
Cough increased (Respiratory, thoracic and mediastinal disorders) | 0/22 | 1/8
Rhinitis (Reproductive system and breast disorders) | 1/22 | 0/8
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3/22 | 0/8
Rash (Skin and subcutaneous tissue disorders) | 1/22 | 0/8
Vesiculobullous rash (Skin and subcutaneous tissue disorders) | 0/22 | 2/8
Abnormal vision (Eye disorders) | 0/22 | 1/8
Ear disorder (Ear and labyrinth disorders) | 1/22 | 0/8
Hematuria (Renal and urinary disorders) | 1/22 | 0/8
Kidney calculus (Renal and urinary disorders) | 1/22 | 0/8
Oliguria (Renal and urinary disorders) | 1/22 | 0/8
Scrotal edema (Renal and urinary disorders) | 0/22 | 1/8
Location reaction to procedure (Injury, poisoning and procedural complications) | 3/22 | 1/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.